CLINICAL TRIAL: NCT05273749
Title: A Phase 3, Double-Blind, Randomized, Multicenter, Placebo-Controlled Study To Evaluate The Efficacy And Safety Of TNX-102 SL Taken Daily At Bedtime In Patients With Fibromyalgia
Brief Title: A Phase 3 Study to Evaluate the Efficacy and Safety of TNX-102 SL Taken Daily in Patients With Fibromyalgia
Acronym: RESILIENT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tonix Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TNX-CY-F307
Record Dates: First submitted 2022-03-01; First posted 2022-03-10 (Actual); Results first posted 2024-12-20 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Fibromyalgia
Keywords: Pain, Sleep, Fibromyalgia, FM
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TNX-102 SL Tablet, 5.6 mg (Experimental): 1 x TNX-102 SL 2.8 mg Tablet taken sublingually each day at bedtime for 2 weeks, then 2 x TNX-102 SL 2.8 mg (5.6 mg) Tablet taken sublingually each day at bedtime for 12 weeks.
  Interventions: Drug: TNX-102 SL Tablet, 5.6 mg
- Placebo SL Tablet (Placebo Comparator): 1 x Placebo Tablet taken sublingually each day at bedtime for 2 weeks, then 2 x Placebo Tablet taken sublingually each day at bedtime for 12 weeks.
  Interventions: Drug: Placebo SL Tablet

INTERVENTIONS:
Drug: TNX-102 SL Tablet, 5.6 mg — Patients will take 1 tablet of randomly assigned study drug sublingually starting on Day 1 for 2 weeks. At the Week 2 visit, all patients will have the dose increased to 2 tablets for 12 weeks.
  Other Names: Low dose cyclobenzaprine sublingual tablets
  Arms: TNX-102 SL Tablet, 5.6 mg
Drug: Placebo SL Tablet — Patients will take 1 tablet of randomly assigned study drug sublingually starting on Day 1 for 2 weeks. At the Week 2 visit, all patients will have the dose increased to 2 tablets for 12 weeks.
  Other Names: Placebo sublingual tablets
  Arms: Placebo SL Tablet

SUMMARY:
This is a Phase 3, randomized, parallel-group, double-blind, placebo-controlled, 14-week study designed to evaluate the efficacy and safety of TNX-102 SL 5.6 mg (2 x 2.8 mg tablets) taken daily at bedtime for the treatment of fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* The patient is male or female 18 to 65 years of age, inclusive.
* The patient has a diagnosis of primary FM as defined by the 2016 Revisions to the 2010/2011 fibromyalgia diagnostic criteria (American College of Rheumatology Preliminary Diagnostic Criteria)

Exclusion Criteria:

* The patient has been diagnosed with infectious or inflammatory arthritis (e.g., rheumatoid arthritis, ankylosing spondylitis, psoriatic arthritis), systemic lupus erythematosus, untreated or active gout (ie, any acute attacks within past 2 years is exclusionary), or meets criteria for other type of systemic autoimmune disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 457 (Actual)
Dates: Start 2022-04-06 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2023-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Sullivan, MD, Study Director — Tonix Pharmaceuticals, Inc.
Locations (33):
- United States (33):
  - Tonix Clinical Site, Phoenix, Arizona
  - Tonix Clinical Site, Oceanside, California
  - Tonix Clinical Site, Santa Ana, California
  - Tonix Clinical Site, Temecula, California
  - Tonix Clinical Site, Cromwell, Connecticut
  - Tonix Clinical Site, Fort Myers, Florida
  - Tonix Clinical Site, Jacksonville, Florida
  - Tonix Clinical Site, Miami Lakes, Florida
  - Tonix Clinical Site, Ocala, Florida
  - Tonix Clinical Site, Oldsmar, Florida
  - Tonix Clinical Site, Orlando, Florida
  - Tonix Clinical Site, Alpharetta, Georgia
  - Tonix Clinical Site, Atlanta, Georgia
  - Tonix Clinical Site, Evansville, Indiana
  - Tonix Clinical Site, West Des Moines, Iowa
  - Tonix Clinical Site, Prairie Village, Kansas
  - Tonix Clinical Site, Covington, Louisiana
  - Tonix Clinical Site, New Orleans, Louisiana
  - Tonix Clinical Site, Prairieville, Louisiana
  - Tonix Clinical Site, Boston, Massachusetts
  - Tonix Clinical Site, Gulfport, Mississippi
  - Tonix Clinical Site, Albuquerque, New Mexico
  - Tonix Clinical Site, Williamsville, New York
  - Tonix Clinical Site, Cincinnati, Ohio
  - Tonix Clinical Site, Tulsa, Oklahoma
  - Tonix Clinical Site, Portland, Oregon
  - Tonix Clinical Site, Charleston, South Carolina
  - Tonix Clinical Site, Austin, Texas
  - Tonix Clinical Site, Dallas, Texas
  - Tonix Clinical Site, McKinney, Texas
  - Tonix Clinical Site, Charlottesville, Virginia
  - Tonix Clinical Site, Danville, Virginia
  - Tonix Clinical Site, Kenosha, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lederman S, Arnold LM, Vaughn B, Engels JM, Kelley M, Sullivan GM. Pain relief by targeting nonrestorative sleep in fibromyalgia: a phase 3 randomized trial of bedtime sublingual cyclobenzaprine. Pain Med. 2026 Jan 1;27(1):86-94. doi: 10.1093/pm/pnaf089. PMID 40627411

RESULTS

PARTICIPANT FLOW:
Groups:
- TNX-102 SL Tablet, 5.6 mg: 1 x TNX-102 SL 2.8 mg Tablet taken sublingually each day at bedtime for 2 weeks, then 2 x TNX-102 SL 2.8 mg (5.6 mg) Tablet taken sublingually each day at bedtime for 12 weeks.
  TNX-102 SL tablet: Patients will take 1 tablet of randomly assigned study drug sublingually starting on Day 1 for 2 weeks. At the Week 2 visit, all patients will have the dose increased to 2 tablets for 12 weeks.
Period: Overall Study
Arm/Group | TNX-102 SL Tablet, 5.6 mg | Placebo SL Tablet
Started | 231 | 226
Completed | 187 | 179
Not Completed | 44 | 47
Not completed — Adverse Event | 14 | 8
Not completed — Lack of Efficacy | 2 | 8
Not completed — Physician Decision | 0 | 2
Not completed — Withdrawal by Subject | 14 | 16
Not completed — Lost to Follow-up | 10 | 10
Not completed — Pregnancy | 1 | 0
Not completed — Non-Compliance | 3 | 2
Not completed — Patient should not have been randomized due to ongoing unstable medical condition | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population: all patients who took investigational product.
Groups:
- TNX-102 SL Tablet, 5.6 mg: 1 x TNX-102 SL 2.8 mg Tablet taken sublingually each day at bedtime for 2 weeks, then 2 x TNX-102 SL 2.8 mg (5.6 mg) Tablet taken sublingually each day at bedtime for 12 weeks.
  TNX-102 SL: Patients will take 1 tablet of randomly assigned study drug sublingually starting on Day 1 for 2 weeks. At the Week 2 visit, all patients will have the dose increased to 2 tablets for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | TNX-102 SL Tablet, 5.6 mg | Placebo SL Tablet | Total
Number analyzed (Participants) | 231 | 226 | 457
Age, Continuous [Mean (Standard Deviation); unit: years] — Patients between the ages of 18-65 at the time of screening were eligible to enroll per protocol entry criteria
  years | 49.3 (10.45) | 49.5 (11.2) | 49.4 (10.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 224 | 212 | 436
  Male | 7 | 14 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 36 | 35 | 71
  Not Hispanic or Latino | 195 | 190 | 385
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 1 | 5 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 32 | 27 | 59
  White | 194 | 192 | 386
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to the Week 14 Endpoint in the Diary NRS Weekly Average of Daily Self Reported Average Pain Severity Scores.
Description: Change from Baseline to the Week 14 endpoint in the diary Numerical Rating Scale (NRS) weekly average of daily self-reported average pain severity scores. Scores range from 0 to 10 where a higher score means worse outcome.
Time Frame: Baseline (Day -7 to Day -1), Week 14
Population: Intention-To-Treat (ITT) population: all patients who were randomized. This is the primary population for efficacy analyses, and patients will be analyzed based on their randomized treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | TNX-102 SL Tablet, 5.6 mg | Placebo SL Tablet
Number analyzed (Participants) | 231 | 225
score on a scale | -1.8 [-2.0 to -1.6] | -1.2 [-1.4 to -0.9]

2. Secondary Outcome: Proportion of Patients With a Patient's Global Impression of Change (PGIC) Rating of "Very Much Improved" or "Much Improved" at the Week 14 Endpoint
Description: The PGIC is a fibromyalgia specific validated instrument on a scale of 1 to 7, where a score of 1 indicates the highest level of improvement and a score of 7 indicates a much worse outcome.
Time Frame: Week 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | TNX-102 SL Tablet, 5.6 mg | Placebo SL Tablet
Number analyzed (Participants) | 231 | 225
Participants | 66 | 34

3. Secondary Outcome: Change From Baseline in the Fibromyalgia Impact Questionnaire - Revised (FIQ-R) Symptoms Domain Score at the Week 14 Endpoint
Description: Change from Baseline in the FIQ-R Symptoms domain score at the Week 14 endpoint. Scores on the symptoms domain range from 0 to 90 where a higher score means worse outcome.
Time Frame: Day 1, Week 14
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | TNX-102 SL Tablet, 5.6 mg | Placebo SL Tablet
Number analyzed (Participants) | 231 | 225
score on a scale | -16.0 [-18.3 to -13.7] | -8.4 [-10.7 to -6.1]

4. Secondary Outcome: Change From Baseline in the FIQ-R Function Domain Score at the Week 14 Endpoint
Description: The FIQ-R is a validated questionnaire. Scores on the function domain range from 0 to 90 where a higher score means worse outcome.
Time Frame: Day 1, Week 14
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | TNX-102 SL Tablet, 5.6 mg | Placebo SL Tablet
Number analyzed (Participants) | 231 | 225
score on a scale | -12.2 [-14.5 to -9.9] | -6.8 [-9.2 to -4.4]

5. Secondary Outcome: Change From Baseline in the Patient Reported Outcomes Measurement Information System (PROMIS) Score for Sleep Disturbance at the Week 14 Endpoint
Description: The PROMIS Sleep disturbance short form 8a consists of 8 questions on a 5-point scale (1 to 5) where a higher score indicates a worse outcome. The total score is reported on a range of 8 to 40. Raw scores are converted to T-scores based on US population with score of 50 as average with a standard deviation of 10.
Time Frame: Day 1, Week 14
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: T-score
Arm/Group | TNX-102 SL Tablet, 5.6 mg | Placebo SL Tablet
Number analyzed (Participants) | 231 | 225
T-score | -8.4 [-9.6 to -7.3] | -4.2 [-5.3 to -3.1]

6. Secondary Outcome: Change From Baseline in the PROMIS Score for Fatigue at the Week 14 Endpoint
Description: The PROMIS fatigue short form 8a consists of 8 questions on a 5 point scale (1 to 5) where a higher score indicates a worse outcome. The total score is reported on a range of 8 to 40. Raw scores are converted to T-scores based on US population with score of 50 as average with a standard deviation of 10.
Time Frame: Day 1, Week 14
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: T-score
Arm/Group | TNX-102 SL Tablet, 5.6 mg | Placebo SL Tablet
Number analyzed (Participants) | 231 | 225
T-score | -7.2 [-8.3 to -6.1] | -4.2 [-5.3 to -3.1]

7. Secondary Outcome: Change From Baseline in the Weekly Average of the Daily Diary Assessment of Sleep Quality at the Week 14 Endpoint
Description: Patients provide a daily numeric assessment of their sleep quality for the previous night, via an electronic diary, using an 11-point NRS. Scores range from 0 (best possible sleep) to 10 (worst possible sleep).
Time Frame: Baseline (Day -7 to Day -1), Week 14
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | TNX-102 SL Tablet, 5.6 mg | Placebo SL Tablet
Number analyzed (Participants) | 231 | 225
score on a scale | -1.8 [-2.0 to -1.5] | -1.2 [-1.4 to -1.0]

ADVERSE EVENTS:
Time Frame: 14 Weeks
Arm/Group | TNX-102 SL Tablet, 5.6 mg | Placebo SL Tablet
All-Cause Mortality (participants affected / at risk) | 0/231 | 0/226
Serious Adverse Events (participants affected / at risk) | 2/231 | 3/226
Other Adverse Events (participants affected / at risk) | 78/231 | 4/226
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TNX-102 SL Tablet, 5.6 mg (N=231) | Placebo SL Tablet (N=226)
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TNX-102 SL Tablet, 5.6 mg (N=231) | Placebo SL Tablet (N=226)
Hypoaesthesia oral (Gastrointestinal disorders) | 55 | 1
Paraesthesia oral (Gastrointestinal disorders) | 16 | 2
Tongue discomfort (Gastrointestinal disorders) | 16 | 0
Product taste abnormal (Product Issues) | 27 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
An industry standard NDA is in place with all study investigators.

DOCUMENTS (2):
  • Study Protocol (2023-06-15): https://cdn.clinicaltrials.gov/large-docs/49/NCT05273749/Prot_002.pdf
  • Statistical Analysis Plan (2023-10-17): https://cdn.clinicaltrials.gov/large-docs/49/NCT05273749/SAP_003.pdf